CLINICAL TRIAL: NCT03847064
Title: Correction of Lower Limb Deformities With Fixator Assisted Nailing
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, shah fahad, RESIDENT, Aga Khan University
Other Study IDs: AKUPK
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Deformity; Bone
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is a retrospective study at a tertiary care hospital. All cases of lower limb deformity whose correction was done with fixator assisted IM nailing from 2010 till 2017 were analyzed.

DETAILED DESCRIPTION:
It is a retrospective study at a tertiary care hospital. All cases of lower limb deformity whose correction was done with fixator assisted IM nailing from 2010 till 2017 were analyzed. Pre Op x-rays and post op x rays will be analyzed for Mechanical Axis Deviation (MAD), anatomical Lateral Distal Femoral Angle (aLDFA), mechanical Lateral Distal Femoral Angle (mLDFA) and Medial Proximal Tibial Angle (MPTA), post-operative activity and functional status of the patients. Data will be analyzed using SPSS

ELIGIBILITY:
Inclusion Criteria:

- All those patients who underwent fixator assisted intramedullary nailing of tibia or femurs for deformity correction were included

Exclusion Criteria:

* Patients who lost to follow up and those with missing records were excluded from the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: .All those patients who has lower limb deformity irrespective of the cause underwent fixator assisted intramedullary nailing of tibia or femurs for deformity correction were included
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Correction of lower limb deformities | 2010 till 2017
  Correction of lower limb deformities with fixator assisted nailing